CLINICAL TRIAL: NCT06339632
Title: Effects of Transcutaneous Electrical Phrenic Nerve Stimulation and Transcutaneous Electrical Diaphragmatic Stimulation: a Randomized Controlled Crossover Trial
Brief Title: Effects of Transcutaneous Electrical Phrenic Nerve Stimulation and Transcutaneous Electrical Diaphragmatic Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AVAP-NG 3363
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Diaphragm
Keywords: Diaphragm; Transcutaneous electrical nerve stimulation; Ultrasound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researchers responsible for assessing diaphragm muscle through ultrasound will perform image recordings and captures during the "TEPNS" and "TEDS" intervention moments. Subsequently, the images will be analyzed by a blinded evaluator for the adopted intervention. The analyses will follow the methods described in the "diaphragm muscle mobility" and "diaphragm muscle thickness and thickening fraction" sections. Study participants will also be instructed not to disclose information regarding their experience and sensations during the intervention period, ensuring study blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous electrical phrenic nerve stimulation (TEPNS) (Experimental): The technique will be performed by applying transcutaneous neuromuscular electrical stimulation to the phrenic nerve pathway in the cervical region.
  Interventions: Other: Transcutaneous electrical phrenic nerve stimulation (TEPNS)
- Transcutaneous electrical diaphragm stimulation (TEDS) (Active Comparator): The technique will be performed by applying transcutaneous neuromuscular electrical stimulation with the electrodes positioned bilaterally in the parasternal region adjacent to the xiphoid process, and the other electrode placed in the intercostal space.
  Interventions: Other: Transcutaneous electrical diaphragm stimulation (TEDS)

INTERVENTIONS:
Other: Transcutaneous electrical phrenic nerve stimulation (TEPNS) — The characteristics of the electrical current: biphasic waves, set at a stimulation frequency of 10 Hz, pulse width of 200 μs, rise time of 1.0 second, on time of 1.0 second, fall time of 1.0 second, and off time of 2 seconds, resulting in 12 stimuli per minute. The application of "TEPNS" will initially be performed by defining the trajectory of the phrenic nerve in the cervical region. The negative pole (active point), a stick with a spherical tip for micro-current of 2 mm will be positioned with slight pressure in the region of the phrenic nerve pathway between the two heads of the sternocleidomastoid muscle. Additionally, at the positive pole (passive point), a self-adhesive electrode sized (2.0 x 2.0 cm) will be positioned on the skin in the shoulder region. The intensity, measured in milliamperes (mA), will be adjusted to the maximum tolerated by the patient. The total stimulation time will be 10 minutes, applied continuously in a single session.
  Arms: Transcutaneous electrical phrenic nerve stimulation (TEPNS)
Other: Transcutaneous electrical diaphragm stimulation (TEDS) — The characteristics of the electrical current are: biphasic waves, set at a stimulation frequency of 30 Hz, pulse width of 400 μs, rise time of 1.0 second, on time of 1.0 second, fall time of 1.0 second, and off time of 2 seconds, resulting in 12 stimuli per minute. Two self-adhesive electrodes sized (5.0 x 5.0 cm) will be used, positioned in the bilateral parasternal region next to the xiphoid process and the other electrode in the intercostal space between the 6th and 7th ribs bilaterally, at the mid-axillary line. The intensity, measured in milliamperes (mA), will be adjusted to the maximum intensity tolerated by the patient until diaphragmatic contraction is observed with the naked eye, without contraction of other muscles in the abdominal region. The total stimulation time will be 10 minutes, applied continuously in a single session.
  Arms: Transcutaneous electrical diaphragm stimulation (TEDS)

SUMMARY:
Transcutaneous electrical phrenic nerve stimulation (TEPNS) and transcutaneous electrical diaphragm stimulation (TEDS) are modalities that use surface electrodes placed on the patients' skin to generate action potentials and contractions of the muscle fibers of the diaphragm. The primary objective will be to evaluate the efficacy of TEPNS and TEDS in healthy adult individuals. Secondary objectives will be to assess the feasibility, safety, and level of discomfort reported by the individual resulting from the application of TEPNS and TEDS.

DETAILED DESCRIPTION:
This crossover trial, single-blind, bicentric study will be conducted at two hospitals. Adult volunteers aged 18 to 60 years, healthy, with a body mass index between 18.5 and 24.9 kg/m2, without a history of previous respiratory diseases, and without contraindications to undergo evaluation or application of the proposed electrical stimulation modalities will be included. Participants' diaphragm muscle will be assessed using ultrasound for variables such as thickness, thickness fraction, and diaphragm mobility. Patients will be randomized using opaque envelope draw prior to evaluation into two distinct experimental moments: 1) "TEPNS" moment - application of the TEPNS protocol; or 2) "TEDS" moment - application of the TEDS protocol. Additionally, data regarding the feasibility and safety of the application of electrical stimulation modalities will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years;
* Normal pulmonary function test, without alterations, assessed through spirometry;
* Body Mass Index (BMI) between 18.5 and 24.9 kg/m2.

Exclusion Criteria:

* Smokers or former smokers;
* Individuals with previously known cardiopulmonary diseases (restrictive lung diseases, chronic obstructive pulmonary disease - COPD, asthma, cystic fibrosis, among other pathologies);
* Presence of implanted electrical devices (pacemaker, implantable cardioverter-defibrillator, among others);
* Individuals who have contraindications to undergo evaluation and/or application of transcutaneous electrical stimulation of the diaphragm muscle, such as: altered sensitivity, wounds at the site of application, deformities, among other conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragm mobility | At baseline, between the fourth and fifth minutes and between the ninth and tenth minutes after the start of stimulation.
  The assessment of diaphragmatic mobility will use a "convex" type transducer (2-6 MHz), positioned in the right subcostal space, at the midclavicular line, tilted in the cephalic direction. The B-mode visualization window will initially be used to locate the diaphragmatic hemi-dome. Upon acquiring a good quality image, respiratory excursions will be measured in M-mode, using the inferior vena cava and the gallbladder as anatomical parameters. Diaphragmatic mobility measurement will be considered as the distance, in centimeters, between the baseline at expiration and its greatest vertical displacement at inspiration produced by diaphragmatic movement.
Diaphragm thickness | At baseline, between the fourth and fifth minutes and between the ninth and tenth minutes after the start of stimulation.
  Diaphragm thickness (Tdi) will be obtained using a high-frequency "linear" type transducer (7-13 MHz), positioned over the zone of apposition (ZA) of the diaphragm muscle. The approximate location is between the 8th and 9th intercostal space, between the anterior axillary line and the midaxillary line, 0.5 to 2.0 cm below the costophrenic angle. The depth will be 1.5 to 3.0 cm, and the diaphragm muscle will be identified as the innermost portion of the hypoechoic muscular layer bounded by two hyperechoic membranes, the pleura - superficial line, and the peritoneum - deeper line. "Tdi" will be measured from the inner edge of the pleural line to the inner edge of the peritoneal line at the end of expiration (Tdi-exp); and at the end of inspiration (Tdi-insp).
Thickening fraction | At baseline, between the fourth and fifth minutes and between the ninth and tenth minutes after the start of stimulation.
  The thickening fraction will be obtained using a high-frequency "linear" type transducer (7-13 MHz), positioned over the zone of apposition (ZA) of the diaphragm muscle. The approximate location is between the 8th and 9th intercostal space, between the anterior axillary line and the midaxillary line, 0.5 to 2.0 cm below the costophrenic angle. The depth will be 1.5 to 3.0 cm, and the diaphragm muscle will be identified as the innermost portion of the hypoechoic muscular layer bounded by two hyperechoic membranes, the pleura - superficial line, and the peritoneum - deeper line. The localization of structures and measurements will be performed in B-mode. The diaphragm thickening fraction will be calculated as the percentage of thickness increment during inspiration relative to the thickness at the end of expiration.

SECONDARY OUTCOMES:
Evaluation of sensory discomfort | At baseline, five and 10 minutes the start of stimulation.
  The assessment of reported sensory discomfort will be measured through the application of the horizontal numerical scale of sensory discomfort. The numerical scale will be presented to participants in its printed version, on standardized paper measuring 10 centimeters in length. The value "0" (zero) will be assigned to the concept of "absence of discomfort," and the value "10" (ten) will be assigned to the concept of "greatest imaginable discomfort."
Safety of TEPNS and TEDS application | The events will be monitored throughout the entire period of TEPNS and TEDS application.
  Safety criteria will be measured through the occurrence of the number of adverse events, including: Mean arterial pressure < 65 mmHg; heart rate > 140 bpm or < 50 bpm; arrhythmias occurrence; oxygen saturation dropping below 88%; temperature increase (above 37.7°C); presence of reported pain above 7 on the visual analog pain scale; presence of burns at the site where electrodes were placed for electrostimulation. The numbers of adverse events will be recorded, along with their classification according to the World Health Organization Patient Safety Document as follows: no harm, minor, moderate, severe, and death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio Libanês, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Boon AJ, Harper CJ, Ghahfarokhi LS, Strommen JA, Watson JC, Sorenson EJ. Two-dimensional ultrasound imaging of the diaphragm: quantitative values in normal subjects. Muscle Nerve. 2013 Jun;47(6):884-9. doi: 10.1002/mus.23702. Epub 2013 Apr 29. PMID 23625789
- [Background] Cancelliero-Gaiad KM, Ike D, Pantoni CB, Mendes RG, Borghi-Silva A, Costa D. Acute effects of transcutaneous electrical diaphragmatic stimulation on respiratory pattern in COPD patients: cross-sectional and comparative clinical trial. Braz J Phys Ther. 2013 Nov-Dec;17(6):547-55. doi: 10.1590/S1413-35552012005000121. Epub 2013 Nov 14. PMID 24271095
- [Background] Canella C, Demondion X, Delebarre A, Moraux A, Cotten H, Cotten A. Anatomical study of phrenic nerve using ultrasound. Eur Radiol. 2010 Mar;20(3):659-65. doi: 10.1007/s00330-009-1579-z. Epub 2009 Sep 2. PMID 19727747
- [Background] Carrillo-Esper R, Perez-Calatayud AA, Arch-Tirado E, Diaz-Carrillo MA, Garrido-Aguirre E, Tapia-Velazco R, Pena-Perez CA, Espinoza-de Los Monteros I, Meza-Marquez JM, Flores-Rivera OI, Zepeda-Mendoza AD, de la Torre-Leon T. Standardization of Sonographic Diaphragm Thickness Evaluations in Healthy Volunteers. Respir Care. 2016 Jul;61(7):920-4. doi: 10.4187/respcare.03999. Epub 2016 Apr 12. PMID 27072012
- [Background] Hedenstierna G, Tokics L, Lundquist H, Andersson T, Strandberg A, Brismar B. Phrenic nerve stimulation during halothane anesthesia. Effects of atelectasis. Anesthesiology. 1994 Apr;80(4):751-60. doi: 10.1097/00000542-199404000-00006. PMID 8024128
- [Background] Santana PV, Cardenas LZ, Albuquerque ALP, Carvalho CRR, Caruso P. Diaphragmatic ultrasound: a review of its methodological aspects and clinical uses. J Bras Pneumol. 2020 Nov 20;46(6):e20200064. doi: 10.36416/1806-3756/e20200064. eCollection 2020. PMID 33237154
- [Background] Testa A, Soldati G, Giannuzzi R, Berardi S, Portale G, Gentiloni Silveri N. Ultrasound M-mode assessment of diaphragmatic kinetics by anterior transverse scanning in healthy subjects. Ultrasound Med Biol. 2011 Jan;37(1):44-52. doi: 10.1016/j.ultrasmedbio.2010.10.004. PMID 21144957